CLINICAL TRIAL: NCT05911698
Title: Fractional co2 Laser Followed by Either Vitamin c or Tranexamic Acid in Treatment of Melasma. Asplit Face Dermoscopic and Clinical Study.
Brief Title: Fractional co2 Laser Followed by Either Vitamin c or Tranexamic Acid in Treatment of Melasma.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Khadija Qenawi (Other)
Responsible Party: Sponsor-Investigator, Khadija Qenawi, Doctor, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fractional laser in melasma
Record Dates: First submitted 2023-03-28; First posted 2023-06-22 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with all types of melasma (Other): Fractional ablative CO2 laser : For each patient, Right side of the face : Fractional ablative CO2 laser will be followed by immediate topical application of vitamin c 3% .
  Left side of the face: Fractional ablative CO2 laser will be followed by immediate topical application of tranexamic acid.
  * Fractional ablative CO2 laser sessions will be performed using the following parameters: power 8-10 W(according to the skin type), spacing 1000 μm (5.3% density), dwell time 400 μs, and stack .
  * During the session, protective goggles will be used both by the patient and by the physician.
  Interventions: Device: Fractional co2 laser

INTERVENTIONS:
Device: Fractional co2 laser — The development of fractional resurfacing has led to improvements to melasma treatment with decreased incidence of post-inflammatory hyperpigmentation; these improvements are due to the enhanced healing times and decreased inflammation as a result of the formation of microscopic columns of tissue destruction.
  These microscopic columns of damaged tissue are surrounded by areas of normal tissue, allowing for shorter migratory paths for the healing keratinocytes.

SUMMARY:
The aim of the study:

1.To compare the efficacy and safety of fractional CO2 laser in combination with vitamin c and tranexamic acid in the treatment of melasma.

2 .To assess the value of dermoscope in measuring of the response to treatment in melasma patients compared to clinical scoring.

DETAILED DESCRIPTION:
Melasma is a chronic dermatologic condition defined by hyperpigmented macules and patches that appear in areas of sun exposure .

Traditionally, the mainstays of treatment for melasma have been topical bleaching agents and strict photoprotection.

Additional adjuvant treatment modalities include chemical peels, dermabrasion, and laser treatments, all of which have demonstrated limited efficacy. There has been an interest in studying the effects of vitamin c and tranexamic acid in melasma.

The development of fractional resurfacing has led to improvements to melasma treatment with decreased incidence of post-inflammatory hyperpigmentation; these improvements are due to the enhanced healing times and decreased inflammation as a result of the formation of microscopic columns of tissue destruction.

These microscopic columns of damaged tissue are surrounded by areas of normal tissue, allowing for shorter migratory paths for the healing keratinocytes.

ELIGIBILITY:
Inclusion Criteria:

1. All types of melasma (epidermal, dermal, and mixed) will be included .
2. Patients older than 19 years of age.

Exclusion Criteria:

1. Pregnancy, breastfeeding.
2. Patients taking drugs that induce facial pigmentation e.g, oral contraceptive pills, or hormonal replacement therapy at the time of the study or during the past 12 months.
3. Patients using of any topical bleaching within 1 month before recruitment.
4. Employment of chemical peels or laser therapy during the past 6 months.
5. Concomitant use of anticoagulants, bleeding disorders.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-10-28 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy and safety of fractional CO2 laser in treatment of melasma. | 1year
  1.: For each patient, Right side of the face : Fractional ablative CO2 laser will be followed by immediate topical application of vitamin c 3% . Left side of the face: Fractional ablative CO2 laser will be followed by immediate topical application of tranexamic acid.
  * Fractional ablative CO2 laser sessions will be performed using the following parameters: power 8-10 W (according to the skin type), spacing 1000 μm (5.3% density), dwell time 400 μs, and stack .
  * During the session, protective goggles will be used both by the patient and by the physician. acid in the treatment of melasma. 2 .To assess the value of dermoscope in measuring of the response to treatment in melasma patients compared to clinical scoring.

CONTACTS AND LOCATIONS:
Overall Officials: Khadija Qenawi, Doctor, Principal Investigator — Assiut University; Hanan Ahmed, Professor, Study Director — Assiut University; Reham Maher, Professor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neeley MR, Pearce FB, Collawn SS. Successful treatment of malar dermal melasma with a fractional ablative CO(2) laser in a patient with type V skin. J Cosmet Laser Ther. 2010 Dec;12(6):258-60. doi: 10.3109/14764172.2010.538412. PMID 21142733
- [Background] Jalaly NY, Valizadeh N, Barikbin B, Yousefi M. Low-power fractional CO(2) laser versus low-fluence Q-switch 1,064 nm Nd:YAG laser for treatment of melasma: a randomized, controlled, split-face study. Am J Clin Dermatol. 2014 Aug;15(4):357-63. doi: 10.1007/s40257-014-0080-x. PMID 24858737
- [Background] Lai D, Zhou S, Cheng S, Liu H, Cui Y. Laser therapy in the treatment of melasma: a systematic review and meta-analysis. Lasers Med Sci. 2022 Jun;37(4):2099-2110. doi: 10.1007/s10103-022-03514-2. Epub 2022 Feb 5. PMID 35122202